CLINICAL TRIAL: NCT03199807
Title: Phase IB/II Study of Personalized New Antigen Reactive Immune Cells (NRT) Combined With Radiotherapy for Advanced Hepatocellular Carcinoma Patients
Brief Title: Phase IB/II Study of NRT Combined With Radiotherapy for Advanced HCC
Acronym: LCRAI-1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Zhengyun Zou, M.D, Ph.D, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nanjing DrumTower Hospital
Record Dates: First submitted 2017-06-18; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: HCC
Keywords: HCC; NRT; TOMO radiotherapy
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: NRT+radiotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NRT + radiotherapy (Experimental): HCC received NRT and radiotherapy
  Interventions: Biological: NRT; Radiation: Radiotherapy

INTERVENTIONS:
Biological: NRT — Peripheral blood lymphocytes will be collected and neoantigen reactive T cells(NRTs) will be generated in the laboratory. NRTs 0.5~1 x 10^10, will be i.v.Q3 weeks for total 4-6 doses.
Radiation: Radiotherapy — Radiotherapy of the major mass by dose of 5Gy/F * 10F

SUMMARY:
The study herein successfully developed a new immunotherapeutic approach combined with radiotherapy, and tried to proved it to be more effective and safe.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common cancer and the third leading cause of cancer-related death worldwide. The resection rate for HCC is approximately 10%-30% and the overall prognosis is very poor with a 5-year survival rate of 5%-6%. The recurrence rate is high after radical resection. In addition to surgery, radiofrequency ablation, transcatheter arterial chemoembolization (TACE), microwave ablation, cryoablation, radioactive seeds implantation, high-intensity-focused ultrasound, radiation therapy, chemotherapy and targeted drugs are available for patients with unresectable tumors; however, the efficacy of these treatments are limited and long-term prognosis in the patients is still poor. Moreover, due to serious side effects induced by treatments such as TACE, chemotherapy and targeted drugs, it may not be possible for patients to continue receiving these therapies. The study herein successfully developed a new immunotherapeutic approach combined with radiotherapy, and tried to proved it to be more effective and safe.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 18 years and over, but no more than 75 years;
2. Histologic or cytologic confirmation of advanced hepatocellular carcinoma;
3. Patients with measurable lesions but can not be treated with surgery;
4. Patients with two or over measurable lesions;
5. ECOG≤0-2, Child-pugh A-B;
6. Patients had not received systemic venous chemotherapy ever before;
7. Hematology Index;
8. Neutrophile granulocyte greater than 1.5×10^9/L;
9. Hemoglobin greater than 10g/dL;
10. Platelet greater than 90×10^9/L;
11. Biochemical index
12. Serum bilirubin not greater than 1.5x upper limit of reference range （ULN）
13. ALT or AST not greater than 1.5x ULN
14. Creatinine clearance no less than 60ml/min;
15. Negative pregnancy test for women of childbearing potential;
16. Provision of informed consent;
17. Be able to follow the research program and follow up process;
18. Expected survival time 3 months or more.

Exclusion Criteria:

1. Chemotherapy with experimental drug within 3 months before the start of study therapy;
2. Have at least another primary malignant tumor;
3. Active infection with bacterial or fungal infection;
4. Patients with HIV infection, HCV infection, serious coronary artery disease or asthma, serious cerebrovascular disease or other diseases that the researchers think can not be entered into the group;
5. Women who are pregnant or breast feeding;
6. Drug abuse, clinical or psychological or social factors which will influence the informed. consent or the study implementation;
7. May be allergic to immunotherapy;
8. Radiotherapy and immunotherapy may not be implemented due to social or geographical factors;
9. Weight loss greater 10% within 6 weeks before the start of study therapy;
10. influence the safety or compliance of the patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-20 (Estimated); Primary Completion 2020-07-20 (Estimated); Study Completion 2021-07-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | up to 6 months
  using Common Terminology Criteria for Adverse Events (CTCAE v4.0) in patients

SECONDARY OUTCOMES:
Response Rate | 3, 6 and 12 months
  Response Rate（RR） will be evaluated according Response Evaluation Criteria
Progression free survival (PFS) | 3, 6, 9 and 12 months
  the duration of progression free survival is measured from the time of treatment to the first date that recurrent or progressive disease or for any reason of death is objectively documented
Overall Survival (OS) | At 6, 12 and 18 months
  the duration is measured from the time of treatment to the time of death

OTHER OUTCOMES:
Th1/Th2 change in the peripheral blood | At baseline,and 1 month, 3 months and 6 months
  cytokines are measured by flow cytometry(FCM)
Interferon-gama change of PBMC cells in the peripheral blood stimulated by tumor antigens | At baseline,and 1 month, 3 months and 6 months
  Interferon-gama change of PBMC cells by ELISPOT

CONTACTS AND LOCATIONS:
Overall Officials: Baorui Liu, M.D & Ph.D, Principal Investigator — The Comprehensive Cancer Centre of Drum Tower Hospital, Medical School of Nanjing University, Clinical Cancer Institute of Nanjing University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu C, Shao J, Dong Y, Xu Q, Zou Z, Chen F, Yan J, Liu J, Li S, Liu B, Shen J. Advanced HCC Patient Benefit From Neoantigen Reactive T Cells Based Immunotherapy: A Case Report. Front Immunol. 2021 Jul 13;12:685126. doi: 10.3389/fimmu.2021.685126. eCollection 2021. PMID 34326839